CLINICAL TRIAL: NCT03986138
Title: Efficacy and Safety of Gadopiclenol for Body Magnetic Resonance Imaging (MRI)
Acronym: PROMISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: GDX-44-011
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Lesion in Body Region
MeSH Terms: interventions — gadopiclenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- gadopiclenol-enhanced MRI then gadobutrol-enhanced MRI (Experimental): Cross-over design: each patient receives gadopiclenol for the first MRI and then gadobutrol for the second MRI
  Interventions: Drug: gadopiclenol; Drug: Gadobutrol 1 MMOLE/ML Intravenous Solution
- gadobutrol-enhanced MRI then gadopiclenol-enhanced MRI (Experimental): Cross-over design: each patient receives gadobutrol for the first MRI and then gadopiclenol for the second MRI
  Interventions: Drug: gadopiclenol; Drug: Gadobutrol 1 MMOLE/ML Intravenous Solution

INTERVENTIONS:
Drug: gadopiclenol — Single intravenous bolus injection
Drug: Gadobutrol 1 MMOLE/ML Intravenous Solution — Single intravenous bolus injection

SUMMARY:
The trial aimed at evaluating the efficacy and the safety of gadopiclenol for body Magnetic resonance Imaging (MRI)

DETAILED DESCRIPTION:
The purpose of this trial was to evaluate a new gadolinium-based contrast agent (GBCA) gadopiclenol in terms of lesion visualization in patients referred for contrast-enhanced MRI of body regions.

This is a prospective, international, multi-center, randomized, double-blind, controlled and cross-over trial.

This trial was conducted in 33 centers worldwide. During the course of the trial, two MRIs were obtained from each patient: one with gadopiclenol and one with gadobutrol. MRI evaluations were assessed by independent off-site blinded readers.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with known or suspected enhancing abnormality(ies) and/or lesion(s) in at least one body region based on a previous imaging procedure performed within 12 months prior to ICF signature. US patients are restricted to the breast in compliance with local approved indications of gadobutrol.

Exclusion Criteria:

* Patient presenting with acute or chronic renal insufficiency, defined as an estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m² assessed within 1 day prior to each contrast agent administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (7):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - UConn Health - University of Connecticut, Farmington, Connecticut
  - The University of Chicago Medical Center, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - University of Missouri Health System, Columbia, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - UT Health San Antonio, San Antonio, Texas
- Acibadem City Clinic Tokuda Hospital Sofia, Sofia, Bulgaria
- France (3):
  - CHU, Angers
  - CHU Beaujon, Clichy
  - Hôpital Saint Louis, Paris
- Germany (4):
  - Klinik für Diagnostische und Interventionelle Radiologie, Aachen
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum des Saarlandes, Homburg
  - University Hospital Jena, Jena
- Hungary (2):
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli, Italy
- Mexico (2):
  - Clinical Research Institute S.C., Estado de México
  - Axis Heilsa S de R.L. de C.V - Althian Clinical Research Management Center, Monterrey
- Poland (5):
  - Szpital Uniwersytecki Nr 1 im. dr Antoniego Jurasza w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Jagiellońskie Centrum Innowacji Sp. z o. o., Krakow
  - Szpital Świętego Rafała, Krakow
  - Centrum Medyczne Affidea Wałbrzych, Wałbrzych
- South Korea (5):
  - Inje University Busan Paik Hospital, Busan
  - Bucheon Suncheonhyang Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Hospital Universitario y Politécnico La Fe, Valencia, Spain
- Ukraine (2):
  - St. Luke's Hospital, Kropyvnytskyi
  - Borys Clinic, Kyiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuhl C, Csoszi T, Piskorski W, Miszalski T, Lee JM, Otto PM. Efficacy and Safety of Half-Dose Gadopiclenol versus Full-Dose Gadobutrol for Contrast-enhanced Body MRI. Radiology. 2023 Jul;308(1):e222612. doi: 10.1148/radiol.222612. PMID 37462494

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among the 324 screened patients,19 were screen failure, 1 received the first contrast agent but was not randomized. A total of 304 patients were randomized, of whom 300 (151 in Arm 1 and 149 in Arm 2) received the first contrast agent and underwent the first MRI (First MRI Period). After a washout period of 2-14 days, 277 patients (141 in the Arm 1 and 136 in the Arm 2) received the second contrast agent and underwent the second MRI (Second MRI Period). 275 patients completed the study.
Groups:
- Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI: Cross-over study design
  For each patient in this Arm, he (she) performed the first contrast-enhanced MRI with gadopiclenol as contrast agent (First MRI Period). After a washout period of 2-14 days (Washout Period), the patient performed the second contrast-enhanced MRI with gadobutrol as contrast agent (Second MRI Period).
  For each patient, two sets of MR images per MRI examination were obtained: unenhanced and gadopiclenol-enhanced MR images obtained in the First MRI Examination Period, unenhanced and gadobutrol-enhanced MR images obtained in the Second MRI Examination Period.
  Gadopiclenol: single intravenous (IV) bolus injection at a rate of 2ml/second
  Gadobutrol 1Mmol/mL Solution for Injection Vial: single intravenous (IV) bolus injection at a rate of 2ml/second
- Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI: Cross-over study design
  For each patient in this Arm, he (she) performed the first contrast-enhanced MRI with gadobutrol as contrast agent (First MRI Period). After a washout period of 2-14 days (Washout Period), the patient performed the second contrast-enhanced MRI with gadopiclenol as contrast agent (Second MRI Period).
  For each patient, two sets of MR images per MRI examination were obtained: unenhanced and gadobutrol-enhanced MR images obtained in the First MRI Examination Period, unenhanced and gadopiclenol-enhanced MR images obtained in the second MRI Examination Period.
  Gadobutrol 1Mmol/mL Solution for Injection Vial: single intravenous (IV) bolus injection at a rate of 2ml/second
  Gadopiclenol: single intravenous (IV) bolus injection at a rate of 2ml/second
Period: First MRI Examination
Arm/Group | Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI | Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI
Started | 152 (A total of 304 patients were randomized before first MRI examination: 152 randomized into Arm 1, for whom gadopiclenol-enhanced MRI had to be performed as First MRI examination, and gadobutrol-enhanced MRI to be performed as Second MRI examination.) | 152 (A total of 304 patients were randomized before first MRI examination: 152 randomized into Arm 2, for whom gadobutrol-enhanced MRI had to be performed as the First MRI examination and gadopiclenol-enhanced MRI to be performed as Second MRI examination.)
Completed | 151 (Among the 152 randomized patients of Arm1, one patients discontinued the trial before receiving the first contrast agent. Therefore, a total of 151 patients of Arm 1 performed the first MRI examination with gadopiclenol as contrast agent.) | 149 (Among the 152 randomized patients of Arm 2, 3 patients discontinued the trial before receiving the first contrast agent. Therefore, a total of 149 patients of Arm 2 performed the first MRI examination with gadobutrol as contrast agent.)
Not Completed | 1 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Other reason (mainly technical issues with MRI machine) | 1 | 2
Period: Washout
Arm/Group | Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI | Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI
Started | 151 | 149
Completed | 141 (Among the 151 patients in the Arm 1 who performed the MRI with gadopiclenol as contrast agent in the First MRI examination Period, 10 patients discontinued the trial before receiving contrast agent (gadobutrol) for the second MRI.) | 136 (Among the 149 patients in the Arm 2 who performed the MRI with gadobutrol as contrast agent in the First MRI examination Period, 13 patients discontinued the trial before receiving contrast agent (gadopiclenol) for the second MRI.)
Not Completed | 10 | 13
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Other reason | 5 | 5
Period: Second MRI Examination
Arm/Group | Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI | Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI
Started | 141 | 136
Completed | 141 (Among the patients in the Arm 1 who performed the MRI with gadopiclenol as contrast agent in the First MRI examination Period, 141 received gadobutrol as contrast agent for the second MRI and completed the study.) | 134 (Among the patients in the Arm 2 who performed the MRI with gadobutrol as contrast agent in the First MRI examination Period, 136 received gadopiclenol as contrast agent for the second MRI. Out of them, 134 completed the study.)
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: The analysis was based on participants. For the primary analysis to demonstrate the superiority of gadopiclenol-enhanced MRI compared to unenhanced MRI, the analysis population was patients who had both Pre (unenhanced) and Paired (combined unenhanced and contrast-enhanced) images with gadopiclenol assessable for primary criteria for at least one matching lesion for at least one off-site reader: 145 patients of Arm 1 who performed first MRI and 133 patients of Arm 2 who performed second MRI.
Groups:
- Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI: Cross-over study design
  For each patient in this Arm, he (she) performed the first contrast-enhanced MRI with gadopiclenol as contrast agent (First MRI Period). After a washout period of 2-14 days (Washout Period), the patient performed the second contrast-enhanced MRI with gadobutrol as contrast agent (Second MRI Period).
  For each patient, two sets of MR images per MRI examination were obtained: unenhanced and gadopiclenol-enhanced MR images obtained in the First MRI Examination Period, unenhanced and gadobutrol-enhanced MR images obtained in the Second MRI Examination Period.
- Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI: Cross-over study design
  For each patient in this Arm, he (she) performed the first contrast-enhanced MRI with gadobutrol as contrast agent (First MRI Period). After a washout period of 2-14 days (Washout Period), the patient performed the second contrast-enhanced MRI with gadopiclenol as contrast agent (Second MRI Period).
  For each patient, two sets of MR images per MRI examination were obtained: unenhanced and gadobutrol-enhanced MR images obtained in the First MRI Examination Period, unenhanced and gadopiclenol-enhanced MR images obtained in the second MRI Examination Period.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI | Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI | Total
Number analyzed (Participants) | 145 | 133 | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.9) | 56.9 (13.1) | 57.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 82 | 164
  Male | 63 | 51 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 20 | 51
  Not Hispanic or Latino | 114 | 113 | 227
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 12 | 30
  Asian | 22 | 22 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 102 | 94 | 196
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 22 | 22 | 44
  Hungary | 28 | 20 | 48
  United States | 27 | 18 | 45
  Ukraine | 4 | 9 | 13
  Poland | 32 | 35 | 67
  Italy | 0 | 1 | 1
  Mexico | 18 | 12 | 30
  France | 8 | 2 | 10
  Bulgaria | 2 | 9 | 11
  Germany | 2 | 3 | 5
  Spain | 2 | 2 | 4
Weight [Mean (Standard Deviation); unit: Kg] | 75.3 (17.1) | 75.5 (17.1) | 75.4 (17.1)

OUTCOME MEASURES:

1. Primary Outcome: Lesion Visualization Comparing Gadopiclenol-enhanced MRI to Unenhanced MRI
Description: The lesion visualization at patient level was based on 3 co-primary criteria on marching lesions: border delineation, internal morphology and degree of contrast enhancement, assessed on the images acquired during the MRI performed with gadopiclenol by 3 independent readers. The independent blinded reader recorded each of the 3 co-primary criteria for up to 3 most representative lesions, using a 4-point scale (1 = poor [internal morphology] or none [border delineation, contrast enhancement], 2 = moderate, 3 = good, 4 = excellent). The mean of scores for each patient and for each co-criterion was calculated as follows: Mean of scores = score of lesion 1 + score of lesion 2 (if any) + score of lesion 3 (if any) divided by the number of lesions, ranged from 1 to 4. The difference in mean scores on matching lesions between Paired [unenhanced and contrast-enhanced] images and Pre-contrast [unenhanced] images was calculated for each of the 3 co-primary criteria and for each reader.
Time Frame: At first MRI examination (gadopiclenol-enhanced MRI) for patients of Arm 1. At second MRI examination (gadopiclenol-enhanced MRI) for patients of Arm 2, performed 2-14 days after gadobutrol-enhanced MRI.
Population: Full Analysis Set (FAS) included a total of 278 patients who had both Pre and Paired images with gadopiclenol assessable for primary criteria for at least one matching lesion for at least one off-site reader: 145 patients in the Arm 1 for whom gadopiclenol-enhanced MRI was performed as first MRI, and 133 patients in the Arm 2 for whom gadopiclenol-enhanced MRI was performed as second MRI. The analysis was based on participants (per patient).
Measure: Least Squares Mean (Standard Error); unit: mean of a score (on a scale) per patient
Groups:
- Patients With Gadopiclenol Paired Images: The analysis included a total of 278 patients on marching lesions who had both gadopiclenol Paired images and gadopiclonol Pre images:
  145 patients of Arm 1 for whom gadopiclenol-enhanced MRI was performed as first MRI, and 133 patients of Arm 2 for whom gadopiclenol-enhanced MRI was performed as second MRI.
  The analysis was based on participants (at patient level).
  Therefore, the 278 patients with gadopiclenol Paired images are the same patients with gadopiclenol Pre images.
- Patients With Gadopiclenol Pre Images: The analysis included a total of 278 patients on marching lesions who had both gadopiclenol Paired images and gadopiclonol Pre images:
  145 patients of Arm 1 for whom gadopiclenol-enhanced MRI was performed as first MRI, and 133 patients of Arm 2 for whom gadopiclenol-enhanced MRI was performed as second MRI.
  The analysis was based on participants (at patient level).
  Therefore, the 278 patients with gadopiclenol Pre images are the same patients with gadopiclenol Paired images.
Arm/Group | Patients With Gadopiclenol Paired Images | Patients With Gadopiclenol Pre Images
Number analyzed (Participants) | 278 | 278
mean of a score (on a scale) per patient
  Border delineation - Reader 1 | 3.79 (0.03) | 2.26 (0.03)
  Border delineation - Reader 2 | 3.48 (0.06) | 3.01 (0.06)
  Border delineation - Reader 3 | 3.49 (0.03) | 1.78 (0.03)
  Internal morphology - Reader 1 | 3.80 (0.02) | 1.99 (0.02)
  Internal morphology - Reader 2 | 3.75 (0.05) | 3.22 (0.05)
  Internal morphology - Reader 3 | 3.72 (0.03) | 1.69 (0.03)
  Contrast enhancement - Reader 1 | 3.64 (0.03) | 1.00 (0.03)
  Contrast enhancement - Reader 2 | 2.82 (0.05) | 1.00 (0.05)
  Contrast enhancement - Reader 3 | 3.33 (0.03) | 1.00 (0.03)
Statistical Analysis 1: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Border delineation; Reader 1. The null hypothesis for primary objective was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error set at 0.025. To conclude the superiority, the null hypothesis had to be rejected for all co-criteria simultaneously and for at least 2 out of 3 readers; Test type: Superiority; p < 0.0001, t-test, 2 sided — To demonstrate the superiority, a statistically significant (one-sided p-value ≤0.025) positive difference in mean scores in border delineation, internal morphology and degree of contrast enhancement of lesions had to be met for 2 out of 3 readers; Mean Difference (Final Values) = 1.53, 95% CI 2-sided [1.46 to 1.60], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Border delineation; Reader 2. The null hypothesis for primary objective was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error set at 0.025. To conclude the superiority, the null hypothesis had to be rejected for all co-criteria simultaneously and for at least 2 out of 3 readers; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [0.36 to 0.58], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Border delineation; Reader 3. The null hypothesis for primary objective was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error set at 0.025. To conclude the superiority, the null hypothesis had to be rejected for all co-criteria simultaneously and for at least 2 out of 3 readers; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.71, 95% CI 2-sided [1.65 to 1.78], Standard Error of Mean 0.04
Statistical Analysis 4: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Internal morphology; Reader 1. The null hypothesis for primary objective was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error set at 0.025. To conclude the superiority, the null hypothesis had to be rejected for all co-criteria simultaneously and for at least 2 out of 3 readers; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.81, 95% CI 2-sided [1.76 to 1.87], Standard Error of Mean 0.03
Statistical Analysis 5: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Internal morphology; Reader 2. The null hypothesis for primary objective was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error set at 0.025. To conclude the superiority, the null hypothesis had to be rejected for all co-criteria simultaneously and for at least 2 out of 3 readers; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [0.42 to 0.64], Standard Error of Mean 0.06
Statistical Analysis 6: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Internal morphology; Reader 3. The null hypothesis for primary objective was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error set at 0.025. To conclude the superiority, the null hypothesis had to be rejected for all co-criteria simultaneously and for at least 2 out of 3 readers; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.03, 95% CI 2-sided [1.95 to 2.11], Standard Error of Mean 0.04
Statistical Analysis 7: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Contrast enhancement; Reader 1. The null hypothesis for primary objective was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error set at 0.025. To conclude the superiority, the null hypothesis had to be rejected for all co-criteria simultaneously and for at least 2 out of 3 readers; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.64, 95% CI 2-sided [2.56 to 2.72], Standard Error of Mean 0.04
Statistical Analysis 8: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Contrast enhancement; Reader 2. The null hypothesis for primary objective was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error set at 0.025. To conclude the superiority, the null hypothesis had to be rejected for all co-criteria simultaneously and for at least 2 out of 3 readers; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.82, 95% CI 2-sided [1.68 to 1.96], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Contrast enhancement; Reader 3. The null hypothesis for primary objective was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error set at 0.025. To conclude the superiority, the null hypothesis had to be rejected for all co-criteria simultaneously and for at least 2 out of 3 readers; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.33, 95% CI 2-sided [2.26 to 2.41], Standard Error of Mean 0.04

2. Secondary Outcome: Lesion Visualization Comparing Gadopiclenol-enhanced MRI to Gadobutrol-enhanced MRI
Description: The lesion visualization (per patient) was based on 3 co-primary criteria: border delineation, internal morphology and degree of contrast enhancement, assessed on the images performed with gadopiclenol and images performed with gadobutrol by 3 independent readers. The independent blinded reader recorded each of the 3 co-primary criteria for up to 3 most representative lesions, using a 4-point scale (1 = poor [internal morphology] or none [border delineation, contrast enhancement], 2 = moderate, 3 = good, 4 = excellent). The mean of scores for each patient and for each of the 3 lesion visualization co-criteria was calculated as follows: Mean of scores = score of lesion 1 + score of lesion 2 (if any) + score of lesion 3 (if any) divided by the number of lesions, ranged from 1 to 4. The difference in mean scores on matching lesions between gadopiclenol scores mean and gadobutrol scores mean was calculated for each of the 3 co-primary criteria and for each reader.
Time Frame: At each of two MRI examinations with an interval of 2-14 days between two MRI examinations
Population: Per-Protocol Set (PPS) analysis including 260 patients (135 patients in the Arm 1 and 125 patients in the Arm 2) with no major protocol deviation who have Paired (combined unenhanced and contrast-enhanced) images for both gadopiclenol and gadobutrol assessable for this secondary outcome mesure for at least one matching lesion for at least one off-site reader. The analysis was based on participants (per patient).
Measure: Least Squares Mean (Standard Error); unit: mean of a score (on a scale) per patient
Groups:
- Patients With Gadopiclenol Paired Images: Analysis included 260 patients with no major protocol deviation who have Paired (combined unenhanced and contrast-enhanced) images for both gadopiclenol and gadobutrol assessable for this secondary outcome mesure for at least one matching lesion for at least one off-site reader: 135 patients of Arm 1 and 125 patients of Arm 2.
  The analysis was based on participants (per patient).
  The 260 patients with gadopiclenol Paired images are the same patients with gadobutrol Paired images.
- Patients With Gadobutrol Paired Images: Analysis included 260 patients with no major protocol deviation who have Paired (combined unenhanced and contrast-enhanced) images for both gadopiclenol and gadobutrol assessable for this secondary outcome mesure for at least one matching lesion for at least one off-site reader: 135 patients of Arm 1 and 125 patients of Arm 2.
  The analysis was based on participants (per patient).
  The 260 patients with gadobutrol Paired images are the same patients with gadopiclenol Paired images.
Arm/Group | Patients With Gadopiclenol Paired Images | Patients With Gadobutrol Paired Images
Number analyzed (Participants) | 260 | 260
mean of a score (on a scale) per patient
  Border delineation - Reader 1 | 3.82 (0.02) | 3.81 (0.02)
  Border delineation - Reader 2 | 3.56 (0.05) | 3.53 (0.05)
  Border delineation - Reader 3 | 3.53 (0.03) | 3.57 (0.03)
  Internal morphology - Reader 1 | 3.83 (0.02) | 3.83 (0.02)
  Internal morphology - Reader 2 | 3.75 (0.04) | 3.75 (0.04)
  Internal morphology - Reader 3 | 3.74 (0.03) | 3.77 (0.03)
  Contrast enhancement - Reader 1 | 3.69 (0.04) | 3.68 (0.04)
  Contrast enhancement - Reader 2 | 2.88 (0.07) | 2.86 (0.07)
  Contrast enhancement - Reader 3 | 3.35 (0.04) | 3.37 (0.04)
Statistical Analysis 1: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Border delineation; Reader 1. The null hypothesis was that the difference in mean scores between gadopiclenol and gadobutrol for each of the 3 primary criteria was equal to the non inferiority margin (-0.35). The alternative hypothesis was that the difference in mean scores between gadopiclenol and gadobutrol for each of the 3 co-primary criteria was greater than the non inferiority margin; Test type: Non-Inferiority — Non-inferiority between gadopiclenol and gadobutrol was concluded if the lower bound of this confidence interval was above the non-inferiority margin set to 0.35 for at least 2 out of 3 blinded readers and for the 3 co-primary criteria simultaneously; p < 0.0001, t-test, 2 sided — The Null hypothesis was rejected if the 2-sided 95% Confidence Interval (CI) for the difference [gadopiclenol scores mean - gadobutrol scores mean] had its lower limit above -0.35; The Student's t-based 95% CIs of the difference between gadopiclenol and gadobutrol were constructed for each of 3 co-primary criteria; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.05 to 0.05], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Border delineation; Reader 2. The null hypothesis was that the difference in mean scores between gadopiclenol and gadobutrol for each of the 3 primary criteria was equal to the non inferiority margin (-0.35). The alternative hypothesis was that the difference in mean scores between gadopiclenol and gadobutrol for each of the 3 co-primary criteria was greater than the non inferiority margin; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.05 to 0.10], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Border delineation; Reader 3. The null hypothesis was that the difference in mean scores between gadopiclenol and gadobutrol for each of the 3 primary criteria was equal to the non inferiority margin (-0.35). The alternative hypothesis was that the difference in mean scores between gadopiclenol and gadobutrol for each of the 3 co-primary criteria was greater than the non inferiority margin; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.10 to 0.01], Standard Error of Mean 0.03
Statistical Analysis 4: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Internal morphology; Reader 1; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.06 to 0.05], Standard Error of Mean 0.03
Statistical Analysis 5: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Internal morphology; Reader 2; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.07 to 0.07], Standard Error of Mean 0.04
Statistical Analysis 6: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Internal morphology; Reader 3; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.08 to 0.02], Standard Error of Mean 0.02
Statistical Analysis 7: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Contrast enhancement; Reader 1; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.06 to 0.09], Standard Error of Mean 0.04
Statistical Analysis 8: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Contrast enhancement; Reader 2; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.07 to 0.12], Standard Error of Mean 0.05
Statistical Analysis 9: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Contrast enhancement; Reader 3; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.08 to 0.04], Standard Error of Mean 0.03

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from informed consent signature up to one day after the second MRI (i.e., minimum of 4 days and a maximum of 23 days)
Groups:
- Gadopiclenol: AEs reported after MRI with gadopiclenol
- Gadobutrol: AEs reported after MRI with gadobutrol
Arm/Group | Gadopiclenol | Gadobutrol
All-Cause Mortality (participants affected / at risk) | 0/288 | 0/290
Serious Adverse Events (participants affected / at risk) | 3/288 | 0/290
Other Adverse Events (participants affected / at risk) | 50/288 | 58/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadopiclenol (N=288) | Gadobutrol (N=290)
Condition Aggravated (General disorders) | 1 (1) | 0 (0) — Not related to contrast-agent or study procedure
Depressed Level Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) — Not related to contrast-agent or study procedure
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) — Not related to contrast-agent or study procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadopiclenol (N=288) | Gadobutrol (N=290)
Injection site pain (General disorders) | 5 (5) | 7 (7)
Injection site bruising (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Injection site discomfort (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Extravasation (General disorders) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 16 (17) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Monocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 2 (2)
Cystatin c increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Paracentesis (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Incorrect dosage administered (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Contrast media reaction (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT03986138/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT03986138/SAP_001.pdf